CLINICAL TRIAL: NCT04570293
Title: The PATCH Trial: Effectiveness and Safety of 5% Lidocaine-medicated Plaster for the Treatment of Trigeminal Neuralgia
Brief Title: 5% Lidocaine-medicated Plaster for the Treatment of Trigeminal Neuralgia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Fang Luo, Director of Department of Pain Management, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KY 2020-102-02
Record Dates: First submitted 2020-09-22; First posted 2020-09-30 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Trigeminal Neuralgia
Keywords: 5% Lidocaine-medicated Plaster; Trigeminal Neuralgia; Enriched Enrollment Randomized Withdrawal; Triggers
MeSH Terms: conditions — Trigeminal Neuralgia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The LMP group (Experimental): The LMP group will receive lidocaine patches (active patches) measuring 10 cm x 14 cm contains 700 mg lidocaine (5% w/w).
  Interventions: Drug: 5% lidocaine medicated plaster
- The control group (Placebo Comparator): The control group will receive vehicle patches that are identical to the active patch, except for the absence of lidocaine, without any optical differences.
  Interventions: Drug: vehicle plaster

INTERVENTIONS:
Drug: 5% lidocaine medicated plaster — The 5% lidocaine medicated plaster is measuring 10 cm x 14 cm contains 700 mg lidocaine (5% w/w) For each patient, the painful area and the trigger point will be chosen for treatment. The investigator will instruct the patient to replace the patch every 12 hours. The patches could be applied during the night (application in the evening and removal in the morning), or during the day. Patients will be told to apply up to three patches at one time.
  Arms: The LMP group
Drug: vehicle plaster — Vehicle patches are identical to the active patch, except for the absence of lidocaine, without any optical differences.For each patient, the painful area and the trigger point will be chosen for treatment. The investigator will instruct the patient to replace the patch every 12 hours. The patches could be applied during the night (application in the evening and removal in the morning), or during the day. Patients will be told to apply up to three patches at one time.
  Arms: The control group

SUMMARY:
Trigeminal neuralgia (TN) is characterized by sudden, severe, usually unilateral, transient, stinging, recurrent electrocute-like shock in one or more divisions of the trigeminal nerve, lasting from a few seconds to less than 2 minutes.Simple daily-life activities, such as washing the face, brushing the teeth, eating, and talking, or the slight touch of trigger points may trigger the attack of pain of TN, resulting in a decline in the patient's quality of life (QoL). Trigger zones predominantly locate in the perioral and nasal region. Paroxysmal pain is associated with triggers in virtually all patients with TN. TN may be caused by abnormality of the trigger zone and the blockade of Na+ channel of trigger zone may be a novel and effective treatment methods for TN. Currently, most patients with TN may not achieve adequate pain relief with a single therapeutic agent. Multiple analgesics targeting different mechanisms of the pain pathway are often used.5% lidocaine medicated plaster (LMP) is a white hydrogel plaster containing adhesive material. LMP was approved for post-herpetic neuralgia (PHN) treatment by the United States Food and Drug Administration (FDA) in 1999. Tamburin et al reported that 2 patients with primary TN who stopped oral drugs because of side effects or refused surgical procedures. Both patients were instructed to wear LMP over the affected area and LMP resulted in reduction of pain intensity and the number of pain paroxysms without side effects. However, due to limitations of these open-label design studies, the observed reductions in pain intensity may have been due to treatment effect, placebo effect, changes in underlying disease state, or a combination of these factors. Therefore, randomized controlled trials will be need to be performed to draw about the efficacy of the LMP in TN.

The PATCH trial is a prospective, double-blinded, vehicle-controlled, parallel-group, multicenter, enriched enrolment with randomized withdrawal (EERW) trial aimed at estimating the efficacy and safety of LMP in patients with TN. After providing informed consent and completing a baseline evaluation, patients will participate in an initial open-label treatment period of LMP (active patches). This openly titrated process is close to clinical practice and can provide data on the proportion of responders and non-responders, the optimal dose of the analgesic drug, and the proportion of withdrawal due to adverse effects. A responder at the end of the open-label treatment phase will be included in the subsequently double-blind treatment phase.

ELIGIBILITY:
Inclusion Criteria:

* Occurrence of episodes of intense facial paroxysmal pain in the distribution(s) of one or more divisions of the trigeminal nerve, triggered by innocuous stimuli;
* Average daily pain intensity ≥ 4 by a brief pain inventory-short form (BPI-SF) Item 5 score (0-10 rating scale of average pain) in the preceding 24-hour period;
* Concomitant analgesic regimens that include 14 days of stable doses with systemic analgesics rather than topical agents for relief of PHN will be permitted
* Normal neurologic examination;
* Normal neuroimaging analysis.

Exclusion Criteria:

* Atypical pain location (eg, no specific trigger points) or trigger zones in the mouth;
* Proposed surgical intervention due to preference of the patient;
* Any condition known to interfere with the correct execution of the sensory tests (eg, peripheral or central neurological dysfunction or cognitive impairments);
* Presence of any other acute or chronic pain disorder with the need of systemic analgesic medication for more than 10 days in the last 3 months;
* Inability to discontinue the use of another lidocaine-containing products or a class I anti-arrhythmic drug during the study period;
* History of hypersensitivity to an amide-type local anesthetic agent, or other contents of the lidocaine or vehicle patch;
* History of surgical intervention or neurological ablation to treatment TN;
* Participation in another clinical trial within 30 days of the study;
* Any patient who was judged to be unreliable or unable to understand the protocol procedures;
* Any abnormality of the skin or of vascular origin at application site;
* Pregnancy or breastfeeding;.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-08-26 (Actual); Study Completion 2022-08-26 (Actual)

PRIMARY OUTCOMES:
the number of treatment failures on LMP vs. number of treatment failures on vehicle patches throughout the double-blind treatment phase | Through study completion, an average of 7 weeks.
  Patients will be defined as treatment failure at the end of the double-blind treatment phase or premature discontinuation if one of the following situations occurs:
  * A 50% or more increase in mean daily pain intensity experienced in the paroxysms within 7-day period of double-blind treatment phase compared to that at the end of initial open-label treatment phase.
  * A 50% or more increase in the total number of paroxysms within 7-day period of double-blind treatment phase compared to that at the end of initial open-label treatment phase.
  * The patient discontinues intervention due to lack of efficacy or intolerable side effects associated study patches.

SECONDARY OUTCOMES:
Time to loss of therapeutic response (LTR) | During the double-blind phase after randomization, an average of 7weeks.
  LTR will be defined as number of days to treatment failure in the double-blind phase after randomization.
Proportion of responders and non-responders | Through the open-label period, an average of 3 weeks.
  A responder at the end of the open-label treatment phase will be defined as follows:
  * A 30% or more decrease in mean daily pain intensity for the 7 days prior to Day 21 compared to that in the baseline phase while the LMP is applied and pain will return or increase when LMP is removed.
  * A 30% or more decrease in the total number of paroxysms for the 7 days prior to Day 21 compared to that in the baseline phase.
  * Regular plaster use will be defined as the plaster are applied every two days.
  * In addition, no intolerable side effects occur at the dose of the existing patch.
the proportion of the patients who report pain relief of 50% or greater | At 3 weeks, 7 weeks
  The pain relief will be assessed by Item 8 on the BPI-SF. Patients will be asked to circle the percentage value from 0% (no relief) to 100% (complete relief) that shows how much pain relief they have achieved during the prior 24 hours at end of open-label phase, and end of double-blind phase or premature discontinuation
The pain intensity | Through study completion, an average of 7 weeks.
  Patients will be asked to circle the number on an 11-point Likert scale of 0 (no pain) to 10 (worst pain imaginable) that describe their worst pain (worst pain), their least pain (least pain) and their pain on average (average pain) in the previous 24 hours and how much pain they are experiencing at the time of the evaluation (pain right now).
The number of paroxysms | Through study completion, an average of 7 weeks.
  The number of paroxysms experienced in the past 4 days weekly
The severity of paroxysms | Through study completion, an average of 7 weeks.
  The severity of paroxysms experienced in the past 4 days weekly
Quality of life (QoL) | Through study completion, an average of 7 weeks.
  Pain interference with the QOL will be assessed by Items 9A-G on the BPI-SF weekly. On these items, patients will be also asked to circle the number on an 11-point Likert scale of 0 (does not interfere) to 10 (completely interferes) that describes the extent to which pain have interfered with their activities of daily living during the prior 24 hours.
Pittsburgh Sleep Quality Index (PSQI) at baseline, at end of open-label phase, and end of double-blind phase or premature discontinuation | At baseline, 3 weeks, 7weeks
  Nineteen individual items generate seven "component" scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The sum of scores for these seven components yields one global score. The total scores are 21. The higher the scores mean the worse the sleep.
Short form 36 health survey questionnaire (SF-36) at baseline, end of open-label phase, and end of double-blind phase or premature discontinuation | At baseline, 3 weeks, 7weeks
  It measures health on eight multi-item dimensions, covering functional status, wellbeing, and overall evaluation of health.
The cost of treatment | Through study completion, an average of 7 weeks.
  The total cost of all medications for TN and the cost of LMP
Patient Global Impression of Change (PGIC) at end of open-label phase, and end of double-blind phase or premature discontinuation | At 3 weeks, 7 weeks
  A 7-point Likert scale, where 1 = very much improved to 7 = very much worse with a value of 4 representing no change
Study blindness | Through study completion, an average of 7 weeks.
  Both the clinician and patient can guess whether the drug used during double-blind phase is LMP or vehicle patches.

CONTACTS AND LOCATIONS:
Overall Officials: Fang Luo, Principal Investigator — Beijing Tiantan Hospital
Locations (5):
- China (5):
  - Beijing Tiantan Hospital, Beijing, Beijing Municipality
  - Beijing China-Janpan Friendship Hospital, Beijing
  - Sanbo Brain Hospital, Capital Medical University, Beijing
  - Jilin province people's hospital, Jilin
  - Linfen People's Hospital, Shanxi

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Background] Di Stefano G, Maarbjerg S, Nurmikko T, Truini A, Cruccu G. Triggering trigeminal neuralgia. Cephalalgia. 2018 May;38(6):1049-1056. doi: 10.1177/0333102417721677. Epub 2017 Jul 14. PMID 28708009
- [Background] Liu M, Zhong J. Mechanism underlying cranial nerve rhizopathy. Med Hypotheses. 2020 Sep;142:109801. doi: 10.1016/j.mehy.2020.109801. Epub 2020 May 6. PMID 32413700
- [Background] Cheville AL, Sloan JA, Northfelt DW, Jillella AP, Wong GY, Bearden Iii JD, Liu H, Schaefer PL, Marchello BT, Christensen BJ, Loprinzi CL. Use of a lidocaine patch in the management of postsurgical neuropathic pain in patients with cancer: a phase III double-blind crossover study (N01CB). Support Care Cancer. 2009 Apr;17(4):451-60. doi: 10.1007/s00520-008-0542-x. Epub 2009 Jan 13. PMID 19142669
- [Background] Gammaitoni AR, Alvarez NA, Galer BS. Safety and tolerability of the lidocaine patch 5%, a targeted peripheral analgesic: a review of the literature. J Clin Pharmacol. 2003 Feb;43(2):111-7. doi: 10.1177/0091270002239817. PMID 12616661
- [Background] Tamburin S, Schweiger V, Magrinelli F, Brugnoli MP, Zanette G, Polati E. Effect of 5% lidocaine medicated plaster on pain intensity and paroxysms in classical trigeminal neuralgia. Ann Pharmacother. 2014 Nov;48(11):1521-4. doi: 10.1177/1060028014544166. Epub 2014 Jul 28. PMID 25070398
- [Derived] Zhao C, Shrestha N, Liu H, Shen Y, Meng L, Fan B, Luo F. The PATCH trial: efficacy and safety of 5% lidocaine-medicated plaster for the treatment of patients with trigeminal neuralgia: a study protocol for a multicentric, double-blind, enriched enrolment randomised withdrawal, vehicle-controlled study. BMJ Open. 2021 Aug 2;11(8):e045493. doi: 10.1136/bmjopen-2020-045493. PMID 34341037